CLINICAL TRIAL: NCT04228731
Title: Cost and Patient Satisfaction Associated With Total Knee Arthroplasty
Brief Title: Inpatient vs Outpatient Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 115081
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Cost; Total Knee Replacement; Outpatient Surgery; Satisfaction; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Personal Satisfaction | interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient (Experimental): Patients in the outpatient group (same day discharge following TKA) are discharged the same day following surgery. All patients are required to meet the discharge criteria to be sent home (i.e., capable of using crutches, relatively free of pain, free of nausea and vomiting, free of excess bleeding, alert and oriented, given take-home medications, and in the company of a caregiver).
  Interventions: Procedure: Outpatient
- Inpatient (Active Comparator): Patients in the inpatient group (following day discharge following TKA) stay in the hospital overnight and then are discharged home the next day. All patients are required to meet the discharge criteria to be sent home (i.e., capable of using crutches, relatively free of pain, free of nausea and vomiting, free of excess bleeding, alert and oriented, given take-home medications, and in the company of a caregiver).
  Interventions: Procedure: Inpatient

INTERVENTIONS:
Procedure: Outpatient — Patients in the outpatient group will be discharged from the hospital the same day of surgery following a total knee arthroplasty
  Arms: Outpatient
Procedure: Inpatient — Patients in the inpatient group will be discharged from the hospital the following day after a total knee arthroplasty
  Arms: Inpatient

SUMMARY:
This is a prospective cohort study comparing standard inpatient (overnight hospital stay) total knee arthroplasty with same day discharge. Patients who are medically well and have a good support structure at home will be recruited. This study will compare patient satisfaction and costs from the perspectives of the Ministry of Health, the institution, society and the patient.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a leading cause of disability and reduced quality of life, presenting a substantial, growing burden to patients and the healthcare system (1). Total knee arthroplasty (TKA) is an established, effective interventions for advanced OA. The prevalence of knee OA is rapidly increasing, resulting in a rising demand for care. The number of procedures is expected to grow by 48%, by 2020 in the US (2). Currently, TKA along with total hip arthroplasty (THA), have a significant impact on healthcare budgets, costing approximately $1.2 billion in annual spending in Canada (3). These staggering numbers highlight the critical need to improve care delivery.

A significant proportion of the overall cost of joint replacement results from the inpatient hospital stay following the procedure. Historically, the standard procedure following TKA required an inpatient hospital stay of two and a half to three weeks, however the introduction of less invasive surgical techniques, improved medical and analgesia management and comprehensive rehabilitation have enabled shorter inpatient stays. Today, the median inpatient stay following TKA is three days in Canada (3). A desire for greater autonomy by the patients as well as patients wanting early mobilization to accelerate recovery and return to activities has led some clinicians to consider an outpatient arthroplasty program. The proposed benefits of outpatient arthroplasty include similar patient outcomes with significantly lower hospital costs, and improved patient satisfaction, independence, and autonomy, however there is a lack of high-quality evidence comparing clinical outcomes of outpatient to inpatient arthroplasty models of care.

A retrospective analysis of over 50,000 THA and TKA procedures found no differences in 30-day major complications or readmissions among patients with a zero to two-day hospital stay compared to those discharged on day three or four postoperative (4). Small cohort studies (5-8) suggest lower costs for outpatients and improved patient satisfaction but have inherent biases; limited to carefully selected patients in privatized health systems.

It is estimated that up to 20% of the overall cost of joint replacement can be attributed to the inpatient stay in hospital at our institution (9). By discharging patients as outpatients, it could be possible to save 20% of the overall costs of joint replacement. Although these preliminary calculations are encouraging, it is not sufficient to effect change solely to achieve cost control, without consideration of safety, effectiveness and patient satisfaction. Further, it is unknown whether the financial savings will be outweighed by additional postoperative costs, increased readmissions or decreased quality of care. A full economic evaluation that simultaneously evaluates cost and effectiveness is crucial prior to implementation. The lack of high-quality evidence regarding its effectiveness warrants a rigorous comparative trial.

The purpose of this study is to evaluate outpatient care pathways for TKA. Specifically, our objectives are to compare the rate of serious adverse events and estimate the cost-effectiveness of outpatient compared to standard inpatient TKA.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee
* Booked for primary unilateral total knee arthroplasty
* Have the ability to read and understand English (printed instructions are provided in English only)
* Home / cell phone access
* Planning to be discharged to home environment
* Patient has an adult to accompany them home post-operatively

Exclusion Criteria:

* Cognitive issues that preclude the ability to understand instructions or provide informed consent
* Lack of a social supports at home
* American Society of Anaesthesiologists (ASA) score equal to or less than 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Indirect and direct costs of treatment | 1 Year
  ER visits, clinician visits, caregiver lost productivity, tests, etc.
Rate of early complications and adverse events | 1 Year
  fall, wound problems, pulmonary embolism, deep vein thrombosis, infection, etc.
Standardized measure of health outcome (EQ-5D) | 1 Year
  utility score measured on a scale of 0 (death) to 1 (perfect health)

SECONDARY OUTCOMES:
Patient satisfaction questionnaire | 2 Weeks
  patient satisfaction with care pre-, peri- and postoperative
Western Ontario McMaster Osteoarthritis Index (WOMAC) | 1 Year
  functional outcome measured on a total scale of 0 (better function) to 100 (worse function) and made up of subscales for pain, stiffness and function
Knee Society Score | 1 Year
  functional outcome measured on a scale of 0 (worse function) to 100 (best function)
Veterans Rand 12 | 1 Year
  quality of life measured on a scale of 0 (worse) to 100 (better) using norm-based scoring
Pain Numeric Rating Scale | 1 Year
  pain measured on a scale from 0 (no pain) to 10 (worst pain imaginable)
Oxford Knee Score - English for Canada | 1 Year
  Level of function, activities of daily living, and effects of pain over preceding four weeks, measured with 12 questions each on a scale from 0 (worst outcome) to 4 (best outcome). A higher score represents a better outcome, with total score range from 1-48.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD, FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz SM, Ong KL, Lau E, Bozic KJ. Impact of the economic downturn on total joint replacement demand in the United States: updated projections to 2021. J Bone Joint Surg Am. 2014 Apr 16;96(8):624-30. doi: 10.2106/JBJS.M.00285. PMID 24740658
- [Background] Sutton JC 3rd, Antoniou J, Epure LM, Huk OL, Zukor DJ, Bergeron SG. Hospital Discharge within 2 Days Following Total Hip or Knee Arthroplasty Does Not Increase Major-Complication and Readmission Rates. J Bone Joint Surg Am. 2016 Sep 7;98(17):1419-28. doi: 10.2106/JBJS.15.01109. PMID 27605685
- [Background] Aynardi M, Post Z, Ong A, Orozco F, Sukin DC. Outpatient surgery as a means of cost reduction in total hip arthroplasty: a case-control study. HSS J. 2014 Oct;10(3):252-5. doi: 10.1007/s11420-014-9401-0. Epub 2014 Jul 12. PMID 25264442
- [Background] Bertin KC. Minimally invasive outpatient total hip arthroplasty: a financial analysis. Clin Orthop Relat Res. 2005 Jun;(435):154-63. doi: 10.1097/01.blo.0000157173.22995.cf. PMID 15930933
- [Background] Lovald ST, Ong KL, Malkani AL, Lau EC, Schmier JK, Kurtz SM, Manley MT. Complications, mortality, and costs for outpatient and short-stay total knee arthroplasty patients in comparison to standard-stay patients. J Arthroplasty. 2014 Mar;29(3):510-5. doi: 10.1016/j.arth.2013.07.020. Epub 2013 Aug 21. PMID 23972298
- [Background] Kolisek FR, McGrath MS, Jessup NM, Monesmith EA, Mont MA. Comparison of outpatient versus inpatient total knee arthroplasty. Clin Orthop Relat Res. 2009 Jun;467(6):1438-42. doi: 10.1007/s11999-009-0730-0. Epub 2009 Feb 18. PMID 19224306
- [Background] Petis SM, Howard JL, Lanting BA, Marsh JD, Vasarhelyi EM. In-Hospital Cost Analysis of Total Hip Arthroplasty: Does Surgical Approach Matter? J Arthroplasty. 2016 Jan;31(1):53-8. doi: 10.1016/j.arth.2015.08.034. Epub 2015 Aug 29. PMID 26387922
- [Background] The Arthritis Alliance of Canada, The Impact of Arthritis in Canada: Today and over the next 30 Years, 2011 http://www.arthritisalliance.ca/en/initiativesen/impact-of-arthritis
- [Background] Canadian Institute for Health Information. Hip and Knee Replacements in Canada, 2017-2018: Canadian Joint Replacement Registry Annual Report. Ottawa, ON: CIHI; 2019.